CLINICAL TRIAL: NCT06669390
Title: A Phase-1b Dose Escalation Study to Assess the Effect of NG11-2 on Radiation Induced Oral Mucositis in Patients With Head & Neck Cancer
Brief Title: A Mouthwash Medicine for the Reduction or Prevention of Mouth Ulceration Caused by Radiotherapy for Head and Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VasoDynamics Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NG11-2-P1b; 2022-002409-99 (EudraCT Number); 87831050 (Other: ISRCTN)
Record Dates: First submitted 2024-10-25; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Oral Mucositis
Keywords: Oral Mucositis; RIOM; Severe Oral Mucositis
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Intervention Model Description: This is an unblinded, single-arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NG11-2 Treatment (Experimental): Patients will undergo daily treatment with NG11-2 immediately prior to radiotherapy for 5 days/week (Mon-Fri) for up to 7 weeks.
  Interventions: Drug: NG11-2

INTERVENTIONS:
Drug: NG11-2 — NG11-2 dose level will vary from 0.92 mg/mL to 5.5 mg/mL during the dose escalation process. The NG11-2 is given as an oral rinse.
  Throughout the radiotherapy regimen, no more than 60 minutes prior to the completion of radiotherapy, on each weekday the patient will rinse their mouth with 12.5 ml of NG11-2 for between 90 & 120 seconds duration, gargling twice for approximately three seconds each if possible during this period then expectorate the solution.

SUMMARY:
This study is looking at a new medication called NG11-2 to see if it can reduce a side effect called severe Radiation-induced Oral Mucositis (RIOM) that can happen to people getting radiation treatment for head and neck cancer. Severe RIOM can make patients very sick and make it hard for them to finish their cancer treatment. Right now, there are no approved drugs that can prevent or treat severe RIOM. This study will test different doses of NG11-2 to find the best one, and then more patients will take that dose to see if it works. This study is being done at multiple hospitals in the UK.

DETAILED DESCRIPTION:
The main objective of the trial is to see if the use of NG11-2, when administered as a mouthwash in head and neck cancer patients prior to their radiotherapy, is tolerable and can reduce or prevent the development of severe radiation induced oral mucositis. More specifically, the trial aims to identify an appropriate dose of NG11-2 IMP based on safety and activity/preliminary efficacy for subsequent assessment in follow-up clinical trials.

Although the primary objective of the trial is to evaluate the safety & tolerability of NG11-2 mouthwash, the secondary objective is to obtain preliminary data on the activity/efficacy of NG11-2 mouthwash in the reduction of severe RIOM.

This is a Phase-1b unblinded, dose escalation, multi-centre study of NG11-2 for the reduction of severe RIOM in Head and Neck cancer patients undergoing radiotherapy, with or without concurrent chemotherapy.

The study design is a "2+4" Dose Escalation design with the following escalation schema (a) If 0 out of 2 enrolled patients have a Dose Limiting Toxicity (DLT) , then escalate to the next Dose Level and enroll 2 more patients (b) if 1 out of 2 patients has a DLT, then add 4 more patients at the same Dose Level (c) if 2 out of 2, or 2 or more out of 6 patients experience a DLT, then stop the dose escalation.

The Maximum Tolerated Dose (MTD) is one dose level below the level at which 2/2 or 2+/6 patients experienced a DLT.

On completion of the Dose Escalation, the Safety Committee will review the available data and a small cohort of patients will be treated at the dose(s) selected by the Safety Committee..

Dosing will start at the 0.92mg/mL (5mM) Dose Level with patients being treated with NG11-2 prior to Radiotherapy on days 1-5 each week for up to 7 weeks.

The proposed patient population for this study includes male and female patients, aged 18 or older with histologically confirmed Head and Neck cancer (preferring oral cavity, oropharyngeal, nasopharyngeal cancer), undergoing primary radical chemoradiotherapy/radiotherapy or adjuvant chemoradiotherapy/radiotherapy with either (a) Extended Oral Cavity, or (b) Buccal Mucosa, or (c) Lips receiving a mean radiation dose of at least 30Gy.

Safety assessments will include evaluation of adverse events (AEs) using NCI CTCAE v5), clinical laboratory assessments (biochemistry, haematology), vital sign measurements (blood pressure, heart rate), 12-lead electrocardiogram (ECG) measurements, and physical examination.

An inspection of the Oral Mucosa will take place every day prior to NG11-2 treatment, except on those days where the Oral Mucositis Scoring Assessment has already occurred, to inspect the condition of the oral mucosa.

The severity of Oral Mucositis (OM) will be scored by trained site staff using WHO, RTOG and NCI-CTCAE v5 scales twice weekly (assessments 72hrs apart) from enrolment to the last study drug treatment, then at weeks 1, 2, 4 and 6 post RT. The WHO scale is the primary scoring scale and the RTOG & NCI-CTCAE v5 scales are exploratory scoring scales.

Additionally, a Patient Reported Outcome Measure - Oral Mucositis (PROM-OM) questionnaire will be performed at each Oral Mucositis Scoring Assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female head and neck cancer patients scheduled for radiotherapy, aged 18 or over on day of signing informed consent;
2. Histologically confirmed head and neck cancer with or without previous resective surgery, having not been previously treated with radiation therapy
3. Scheduled to receive a mean radiation dose of no less than 30 Gy on either (a) Extended Oral Cavity, or (b) Buccal Mucosa, or (c) Lips, according to CT-based delineation of Organ-At-Risk (OAR) Guideline, with or without concurrent chemotherapy (Section 13.8 for guidance);
4. Rendered dentally fit for radiotherapy;
5. Have a Performance Status >60 on the Karnofsky scale
6. No evidence of active systemic infections at the time of screening;
7. No oral fungal infection by visual examination or swab test;
8. Body Mass Index >=18.5 kg/m²
9. Normalcy of diet evaluated with the Performance Status Scale for Head and Neck cancer patients (PSSHN) >=30;
10. Ability to retain and swill liquid inside the oral cavity for at least 90 seconds;
11. Female patients of childbearing potential must have a negative urine or serum pregnancy test during the 2 week Screening period
12. Provide written informed consent for the trial.
13. Consent to utilize medically acceptable methods of contraception throughout the study period if of child-bearing potential;
14. Be able to comply with protocol procedures (such as Oral Mucositis assessment and swish/spit) and study schedule

Exclusion Criteria:

1. Tumour of the larynx
2. Mentally or legally incapacitated, in the opinion of the PI, which could interfere with the ability of the patient to understand or adhere to the requirements of the study;
3. Open or unhealed non-cancerous wounds or ulcers in the oral cavity;
4. WHO Oral Mucositis grade of 2 or more
5. Uncontrolled Hypertension, defined as blood pressure in adults >150/100mm Hg at screening;
6. A known clinically significant abnormal ECG, such as arrhythmia and active ischemia,within 6 months prior to treatment;
7. Xerostomia or hyposalivation;
8. Known allergy or intolerance to sympathomimetic drugs (e.g., pseudoephedrine, epinephrine), alcohol, or any NG11-2 excipient;
9. Receiving monoamine oxidase (MAO) inhibitors or antidepressants (triptyline or imipramine types); Use of MAO inhibitor in the 14 days prior to treatment, such as isocarboxazid, linezolid, methylene blue injection, phenelzine, rasagiline, selegiline, or tranylcypromine;
10. History or current evidence of clinically significant laboratory abnormality or any disease condition that might confound the results of the study, or interfere with the patient's participation for the full duration of the study
11. Current participation in any other oral mucositis studies or completion/ withdrawal from any other oral mucositis studies within the last 3 months
12. Patient is, at the time of signing informed consent, a regular user of any illicit drugs, which would interfere with cooperation with the requirements of the trial;
13. Patient is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study;
14. Any other condition which, in the opinion of the Investigator, means that the patient is not a good candidate for study enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Occurence of Dose Limiting Toxicities (DLT) | Dose Limiting Toxicities will be evaluated throughout the study from time of patient consent until 42 days after last IMP dose
Occurence of Serious Adverse Events (SAE) | Serious Adverse Events will be evaluated throughout the study from time of patient consent until 42 days after last IMP dose

SECONDARY OUTCOMES:
Duration of severe Radiation-Induced Oral Mucositis (World Health Organisation Grade 0-4, higher = worse) | From screening and twice weekly in each week of study treatment and then at up to 42 days post end of Radiotherapy, in the follow-up period.
Duration of severe Radiation-Induced Oral Mucositis (Radiation Therapy Oncology Group Grade 0-4, higher = worse) | From screening and twice weekly in each week of study treatment and then at up to 42 days post end of Radiotherapy, in the follow-up period.
Duration of severe Radiation-Induced Oral Mucositis (National Cancer Institute - Common Toxicity Criteria for Adverse Events V5 Grade 1-5, higher = worse) | From screening and twice weekly in each week of study treatment and then at up to 42 days post end of Radiotherapy, in the follow-up period.
Incidence of severe Radiation-Induced Oral Mucositis (World Health Organisation Grade 0-4, higher = worse | From screening and twice weekly in each week of study treatment and then at up to 42 days post end of Radiotherapy, in the follow-up period.
Incidence of severe Radiation-Induced Oral Mucositis (Radiation Therapy Oncology Group Grade 0-4, higher = worse) | From screening and twice weekly in each week of study treatment and then at up to 42 days post end of Radiotherapy, in the follow-up period.
Incidence of severe Radiation-Induced Oral Mucositis (National Cancer Institute - Common Toxicity Criteria for Adverse Events V5 Grade 1-5, higher = worse) | From screening and twice weekly in each week of study treatment and then at up to 42 days post end of Radiotherapy, in the follow-up period.
Time to onset of severe Radiation-Induced Oral Mucositis (World Health Organisation Grade 0-4, higher = worse | From screening and twice weekly in each week of study treatment and then at up to 42 days post end of Radiotherapy, in the follow-up period.
Time to onset of severe Radiation-Induced Oral Mucositis (Radiation Therapy Oncology Group Grade 0-4, higher = worse) | From screening and twice weekly in each week of study treatment and then at up to 42 days post end of Radiotherapy, in the follow-up period.
Time to Onset of severe Radiation-Induced Oral Mucositis (National Cancer Institute - Common Toxicity Criteria for Adverse Events V5 Grade 1-5, higher = worse) | From screening and twice weekly in each week of study treatment and then at up to 42 days post end of Radiotherapy, in the follow-up period.
Impact of Oral Mucositis on patient's oral pain and ability to eat and drink | From screening and twice weekly in each week of study treatment and then at up to 42 days post end of Radiotherapy, in the follow-up period.
  Patient Reported Outcome Measure - Oral Mucositis (PROM-OM)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Mary Lei, Principal Investigator — Guy's & St Thomas' Hospital
Locations (4):
- United Kingdom (4):
  - Aberdeen Royal Infirmary, Aberdeen
  - Belfast City Hospital, Belfast
  - Queen Elizabeth Hospital, Birmingham
  - Guy's & St Thomas' Hospital, London